CLINICAL TRIAL: NCT02120573
Title: Evaluation of Teaching Methods in Mass CPR Training in Different Groups of the Society
Brief Title: Efficacy of CPR Teaching in Mass Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shiraz education development center (Unknown)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 93-1345
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Teaching CPR
Keywords: Cardiac Arrest; Cardiopulmonary Resuscitation; Training
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- medical students (Active Comparator): medical students took part in workshop
  Interventions: Other: Workshop using Lecture and human model; Other: Workshop using Educational Film; Other: Workshop using Lecture, human model as well as Educational Film; Other: Workshop using Lecture, human model, Educational Film as well as reference book
- general population (Active Comparator): general population took part in workshop
  Interventions: Other: Workshop using Lecture and human model; Other: Workshop using Educational Film; Other: Workshop using Lecture, human model as well as Educational Film; Other: Workshop using Lecture, human model, Educational Film as well as reference book
- nonmedical students (Active Comparator): all students from different subjects, non medical and paramedical
  Interventions: Other: Workshop using Lecture and human model; Other: Workshop using Educational Film; Other: Workshop using Lecture, human model as well as Educational Film; Other: Workshop using Lecture, human model, Educational Film as well as reference book

INTERVENTIONS:
Other: Workshop using Lecture and human model — workshop to teach CPR with lecture and human models
Other: Workshop using Educational Film — workshops using film review about CPR
Other: Workshop using Lecture, human model as well as Educational Film — using educational films and human model and lecture for training
Other: Workshop using Lecture, human model, Educational Film as well as reference book — training volunteers with lecture, films, and human models and giving them reference book for referral

SUMMARY:
This prospective study evaluate teaching efficacy of CPR training using different methods in general population, medical students and non medical students with the 12 months evaluation of its recall

DETAILED DESCRIPTION:
In a prospective and observational study of 2000 individuals in three different groups including medical students, non-medical students and general populations four different protocols of CPR training were applied and their efficacy were compared between the groups. Meanwhile, 12 months after the study course, 460 participants from three groups were asked to take part in a theoretical and practical exam to evaluate the long term efficacy of the four protocols.

ELIGIBILITY:
Inclusion Criteria:

* all participant take part in workshop

Exclusion Criteria:

* refuse to take part in exams

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
teaching efficacy | 24 hours
  pre test and post test exam before and after workshop
late post workshop practical test | 12 months
  practical exam about general measures of CPR

SECONDARY OUTCOMES:
trainee satisfaction | 24 hours
  questionaire showing their satisfaction about the workshop

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciencs, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Hasani H, Bahrami M, Malekpour A, Dehghani M, Allahyary E, Amini M, Abdorahimi M, Khani S, Kalantari Meibodi M, Kojuri J. Evaluation of Teaching Methods in Mass CPCR Training in Different Groups of the Society, an Observational Study. Medicine (Baltimore). 2015 May;94(21):e859. doi: 10.1097/MD.0000000000000859. PMID 26020392